CLINICAL TRIAL: NCT01235338
Title: A Phase 1, Open-label, Drug Interaction Study Evaluating the Pharmacokinetic Profiles of SPD489 and EFFEXOR XR, Administered Alone and in Combination in Healthy Adult Subjects
Brief Title: Co-Administration of LDX (SPD489) and Venlafaxine XR (EFFEXOR XR) in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SPD489-117
Record Dates: First submitted 2010-11-02; First posted 2010-11-05 (Estimated); Results first posted 2011-12-08 (Estimated); Last update posted 2021-06-14 (Actual); Status verified 2021-06

CONDITIONS: Healthy
MeSH Terms: interventions — Lisdexamfetamine Dimesylate; Venlafaxine Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- LDX (SPD489) + Venlafaxine XR (Effexor XR) (Experimental)
  Interventions: Drug: LDX + Venlafaxine XR
- Venlafaxine XR + LDX (Experimental)
  Interventions: Drug: Venlafaxine XR + LDX

INTERVENTIONS:
Drug: LDX + Venlafaxine XR — * Day 1-5 LDX 30mg
  * Day 6-10 LDX 50mg
  * Day 11-15 LDX 70mg
  * Day 16-20 LDX 70mg and Venlafaxine XR 75mg daily
  * Day 21-25 LDX 70mg and Venlafaxine XR 150mg daily
  * Day 26-30 LDX 70mg and Venlafaxine XR 225mg daily
  * Day 31-34 Venlafaxine XR 150mg daily
  * Day 35-38 Venlafaxine XR 75mg daily.
  Other Names: Lisdexamfetamine dimesylate, LDX, Vyvanse, SPD489; Venlafaxine hydrochloride extended-release, Effexor XR,
  Arms: LDX (SPD489) + Venlafaxine XR (Effexor XR)
Drug: Venlafaxine XR + LDX — * Day 1-5 Venlafaxine XR 75mg
  * Day 6-10 Venlafaxine XR 150mg
  * Day 11-15 Venlafaxine XR 225mg
  * Day 16-20 Venlafaxine XR 225mg and LDX 30mg daily
  * Day 21-25 Venlafaxine XR and LDX 50mg daily
  * Day 26-30 Venlafaxine XR 225mg and LDX 70mg daily
  * Day 31-34 Venlafaxine XR 150mg
  * Day 35-38 Venlafaxine XR 75mg.
  Other Names: Venlafaxine hydrochloride extended-release, Effexor XR; Lisdexamfetamine dimesylate, LDX, Vyvanse, SPD489
  Arms: Venlafaxine XR + LDX

SUMMARY:
This study will examine the effects of co-administration of SPD489 and the antidepressant EFFEXOR XR on the pharmacokinetics of lisdexamfetamine, d-amphetamine, and EFFEXOR XR. In addition, serial blood pressure and pulse measures will be obtained and examined to ensure that there are no unexpected changes in vital signs following co administration of SPD489 and EFFEXOR XR that would impact the further study of this drug combination. The hypothesis is that a drug drug interaction could possibly exist.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-45 years
2. Subject is willing to comply with any applicable contraceptive requirements of the protocol and is:

   * Male, or
   * Non-pregnant, non-lactating female
   * Females must be at least 90 days post partum or nulliparous.
3. Female subjects must have a negative serum beta Human Chorionic Gonadotropin (HCG) pregnancy test
4. Satisfactory medical assessment
5. Ability to provide information on family history of hypertension.
6. Body Mass Index (BMI) between 18.5 and 30.0kg/m² inclusive.
7. Ability to swallow all investigational products.

Exclusion Criteria:

1. Current or recurrent disease (e.g., cardiovascular, renal, liver, gastrointestinal, malignancy or other conditions)
2. Current or relevant previous history of physical or psychiatric illness.
3. Significant illness.
4. History of significant anxiety, tension, or agitation as assessed by the Investigator.
5. History of or current diagnosis of glaucoma.
6. History of a seizure disorder (other than infantile febrile seizures), any tic disorder or a current diagnosis and/or known family history of Tourette's Disorder.
7. History of symptomatic cardiovascular disease, advanced arteriosclerosis, structural cardiac abnormality, cardiomyopathy, serious heart rhythm abnormalities, coronary artery disease, transient ischemic attack or stroke, or other serious cardiac problems.
8. History of controlled or uncontrolled hypertension or a resting sitting systolic BP >139mmHg or diastolic BP >89mmHg.
9. Known family history of sudden cardiac death or ventricular arrhythmia.
10. Suicidal ideation or any lifetime history of suicidal behavior.
11. Consumption of alcohol, Seville oranges, grapefruit, or any grapefruit containing products within 7 days of first dose of investigational product.
12. Current use of any medication (including prescription, over the counter [OTC], herbal or homeopathic preparations or supplements) with the exception of the occasional dose of acetaminophen, or hormonal contraceptives.
13. History of alcohol or other substance abuse within the last year.
14. A positive screen for alcohol or drugs of abuse.
15. Male subjects who consume more than 21 units of alcohol per week or 3 units per day. Female subjects who consume more than 14 units of alcohol per week or 2 units per day. [1 alcohol unit =1 beer = 1 wine (5oz) = 1 liquor (1.5oz) = 0.75oz alcohol]
16. A positive human immunodeficiency virus (HIV) antibody screen, Hepatitis B surface antigen (HBsAg), or Hepatitis C virus (HCV) antibody screen.
17. Use of tobacco in any form (e.g., smoking or chewing) or other nicotine-containing products in any form (e.g. gum, patch). Ex-users must report that they have stopped using tobacco for at least 30 days prior to receiving the first dose of investigational product.
18. Routine consumption of more than 2 units of caffeine per day or subjects who experience caffeine withdrawal headaches. (One caffeine unit is contained in the following items: one 6oz. cup of coffee, two 12oz. cans of cola, one 12oz. cup of tea, three 1oz. chocolate bars, or one 8oz. serving of an energy drink. Decaffeinated coffee, tea, or cola are not considered to contain caffeine).
19. Donation of blood or blood products (e.g., plasma or platelets) within 60 days prior to receiving the first dose of investigational product.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2010-10-28 (Actual); Primary Completion 2010-12-30 (Actual); Study Completion 2011-01-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (1):
- Clinical Pharmacology of Miami, Miami, Florida, United States

REFERENCES:
- [Result] Ermer J, Haffey MB, Richards C, Lasseter K, Roesch B, Purkayastha J, Corcoran M, Harlin B, Martin P. An open-label investigation of the pharmacokinetic profiles of lisdexamfetamine dimesylate and venlafaxine extended-release, administered alone and in combination, in healthy adults. Clin Drug Investig. 2013 Apr;33(4):243-54. doi: 10.1007/s40261-013-0073-1. PMID 23512639
- See also: FDA Recall Information — http://www.fda.gov/opacom/7alerts.html

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of the 80 randomized subjects, 3 did not receive any investigational product and therefore were not included in the Safety Analysis/Pharmacokinetic Analysis Sets (n = 77).
Groups:
- LDX + Venlafaxine XR: LDX (Lisdexamfetamine Dimesylate, SPD489, Vyvanse®) 30 mg once daily (QD) Days 1-5, then LDX 50 mg QD Days 6-10, then LDX 70 mg QD Days 11-15, then LDX 70 mg + venlafaxine XR (Venlafaxine Hydrochloride extended-release, Effexor® XR) 75 mg QD Days 16-20, then LDX 70 mg + venlafaxine XR 150 mg QD Days 21-25, then LDX 70 mg + venlafaxine XR 225 mg QD Days 26-30, then venlafaxine XR 150 mg QD Days 31-34, then venlafaxine XR 75 mg QD Days 35-38.
- Venlafaxine XR + LDX: Venlafaxine XR (Venlafaxine Hydrochloride extended-release, Effexor® XR) 75 mg QD Days 1-5, then venlafaxine XR 150 mg QD Days 6-10, then venlafaxine XR 225 mg QD Days 11-15, then venlafaxine XR 225 mg + LDX (Lisdexamfetamine Dimesylate, SPD489, Vyvanse®) 30 mg QD Days 16-20, then venlafaxine XR 225 mg + LDX 50 mg QD Days 21-25, then venlafaxine XR 225 mg + LDX 70 mg QD Days 26-30, then venlafaxine XR 150 mg QD Days 31-34, then venlafaxine XR 75 mg QD Days 35-38.
Period: Overall Study
Arm/Group | LDX + Venlafaxine XR | Venlafaxine XR + LDX
Started | 42 | 38
Completed | 31 | 33
Not Completed | 11 | 5
Not completed — Adverse Event | 3 | 2
Not completed — Protocol Violation | 1 | 1
Not completed — Withdrawal by Subject | 5 | 0
Not completed — Exclusion criteria violations | 1 | 1
Not completed — Positive drug screen | 0 | 1
Not completed — Prohibited meds | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | LDX + Venlafaxine XR | Venlafaxine XR + LDX | Total
Number analyzed (Participants) | 40 | 37 | 77
Age, Continuous [Mean (Standard Deviation); unit: years] — The Safety Analysis Set (n = 77) was used to calculate Baseline Measures. The Safety Analysis Set is defined as all enrolled subjects who took at least 1 dose of investigational product and had at least 1 post-dose safety assessment. 80 subjects were enrolled but 3 never received investigational product.
  years | 33.2 (7.01) | 33.8 (7.29) | 33.5 (7.10)
Age, Customized [Count of Participants; unit: Participants]
  Between 18 and 45 years | 40 | 37 | 77
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 10 | 22
  Male | 28 | 27 | 55
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 40 | 37 | 77

OUTCOME MEASURES:

1. Primary Outcome: Maximum Plasma Concentration (Cmax) of Lisdexamfetamine Dimesylate
Description: Lisdexamfetamine dimesylate (SPD489) itself is inactive, but following oral administration is converted to the active isomer, d-amphetamine, that is responsible for the drug's therapeutic activity.
Time Frame: Day 15 and Day 30 (24 hour sampling)
Population: Pharmacokinetic Analysis Set (PAS) defined as all subjects who took a t least 1 dose of investigational product and had at least 1 post-dose safety assessment and who had no major deviations related to investigational product intake (e.g. vomiting) and for whom the primary pharmacokinetic data were considered sufficient and interpretable.
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | LDX + Venlafaxine XR | Venlafaxine XR + LDX
Number analyzed (Participants) | 32 | 34
ng/ml
  Day 15 | 49.06 (32.25) | 0 (0)
  Day 30 | 49.84 (34.3) | 50.77 (19.68)

2. Primary Outcome: Cmax of d-Amphetamine
Description: d-Amphetamine is the active isomer of Lisdexamfetamine dimesylate (SPD489) and is responsible for the drug's therapeutic activity.
Time Frame: Day 15 and Day 30 (24 hour sampling)
Population: PAS
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | LDX + Venlafaxine XR | Venlafaxine XR + LDX
Number analyzed (Participants) | 32 | 34
ng/ml
  Day 15 | 88.91 (26.87) | 0 (0)
  Day 30 | 88.91 (22.72) | 85.27 (20.55)

3. Primary Outcome: Cmax of Venlafaxine Hydrochloride
Description: Venlafaxine Hydrochloride is the active ingredient of Effexor XR
Time Frame: Day 15 and Day 30 (24 hour sampling)
Population: PAS
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | LDX + Venlafaxine XR | Venlafaxine XR + LDX
Number analyzed (Participants) | 32 | 34
ng/ml
  Day 15 | 0 (0) | 210.98 (120.6)
  Day 30 | 198.5 (105.48) | 228.89 (124.42)

4. Secondary Outcome: Systolic Blood Pressure
Time Frame: Baseline and up to 39 days
Population: Safety Analysis Set (SAS) defined as all enrolled subjects who took at least 1 dose of investigational product and had at least 1 post-dose safety assessment.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | LDX + Venlafaxine XR | Venlafaxine XR + LDX
Number analyzed (Participants) | 40 | 37
mmHg
  Baseline | 110.17 (8.996) | 110.48 (9.623)
  Up to 39 Days | 117.82 (8.547) | 121.51 (7.695)

5. Secondary Outcome: Diastolic Blood Pressure
Time Frame: Baseline and up to 39 days
Population: SAS
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | LDX + Venlafaxine XR | Venlafaxine XR + LDX
Number analyzed (Participants) | 40 | 37
mmHg
  Baseline | 73.69 (7.446) | 73.68 (6.730)
  Up to 39 Days | 77.85 (6.628) | 80.45 (7.4515)

6. Primary Outcome: Cmax of o-Desmethylvenlafaxine
Description: Venlafaxine, after oral administration, is metabolized in the liver to an active metabolite, o-Desmethylvenlafaxine.
Time Frame: Day 15 and Day 30 (24 hour sampling)
Population: PAS
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | LDX + Venlafaxine XR | Venlafaxine XR + LDX
Number analyzed (Participants) | 32 | 34
ng/ml
  Day 15 | 0 (0) | 420.55 (139.67)
  Day 30 | 413.71 (149.97) | 371.54 (104.92)

7. Primary Outcome: Cmax of Composite (Venlafaxine + o-Desmethylvenlafaxine)
Time Frame: Day 15 and Day 30 (24 hour sampling)
Population: PAS
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | LDX + Venlafaxine XR | Venlafaxine XR + LDX
Number analyzed (Participants) | 32 | 34
ng/ml
  Day 15 | 0 (0) | 624.56 (179.7)
  Day 30 | 603.49 (181.32) | 588.68 (158.79)

8. Primary Outcome: Area Under the Steady-state Plasma Concentration-time Curve (AUC) of Lisdexamfetamine Dimesylate
Time Frame: Day 15 and Day 30 (24 hour sampling)
Population: PAS
Measure: Mean (Standard Deviation); unit: ng*hr/ml
Arm/Group | LDX + Venlafaxine XR | Venlafaxine XR + LDX
Number analyzed (Participants) | 32 | 34
ng*hr/ml
  Day 15 | 65.5 (44.0) | 0 (0)
  Day 30 | 63.9 (43.7) | 60.8 (19.2)

9. Primary Outcome: AUC of d-Amphetamine
Time Frame: Day 15 and Day 30 (24 hour sampling)
Population: PAS
Measure: Mean (Standard Deviation); unit: ng*hr/ml
Arm/Group | LDX + Venlafaxine XR | Venlafaxine XR + LDX
Number analyzed (Participants) | 32 | 34
ng*hr/ml
  Day 15 | 1143.4 (292.8) | 0 (0)
  Day 30 | 1135.4 (301.5) | 1049.2 (268.7)

10. Primary Outcome: AUC of Venlafaxine Hydrochloride
Time Frame: Day 15 and Day 30 (24 hour sampling)
Population: PAS
Measure: Mean (Standard Deviation); unit: ng*hr/ml
Arm/Group | LDX + Venlafaxine XR | Venlafaxine XR + LDX
Number analyzed (Participants) | 32 | 34
ng*hr/ml
  Day 15 | 0 (0) | 2900.0 (1919.3)
  Day 30 | 2839.7 (1706.8) | 3202.6 (1942.5)

11. Primary Outcome: AUC of o-Desmethylvenlafaxine
Time Frame: Day 15 and Day 30 (24 hour sampling)
Population: PAS
Measure: Mean (Standard Deviation); unit: ng*hr/ml
Arm/Group | LDX + Venlafaxine XR | Venlafaxine XR + LDX
Number analyzed (Participants) | 32 | 34
ng*hr/ml
  Day 15 | 0 (0) | 8363.3 (2168.1)
  Day 30 | 8061.3 (2868.7) | 6955.1 (1962.8)

12. Primary Outcome: AUC of Composite (Venlafaxine + o-Desmethylvenlafaxine)
Time Frame: Day 15 and Day 30 (24 hour sampling)
Population: PAS
Measure: Mean (Standard Deviation); unit: ng*hr/ml
Arm/Group | LDX + Venlafaxine XR | Venlafaxine XR + LDX
Number analyzed (Participants) | 32 | 34
ng*hr/ml
  Day 15 | 0 (0) | 10738.0 (3273.3)
  Day 30 | 10673.9 (3035.7) | 10342.2 (3096.1)

13. Primary Outcome: Time of Maximum Plasma Concentration (Tmax) of Lisdexamfetamine Dimesylate
Time Frame: Day 15 and Day 30 (24 hour sampling)
Population: PAS
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | LDX + Venlafaxine XR | Venlafaxine XR + LDX
Number analyzed (Participants) | 32 | 34
hours
  Day 15 | 1.1 (0.3) | 0 (0)
  Day 30 | 1.1 (0.3) | 1.0 (0.3)

14. Primary Outcome: Tmax of d-Amphetamine
Time Frame: Day 15 and Day 30 (24 hour sampling)
Population: PAS
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | LDX + Venlafaxine XR | Venlafaxine XR + LDX
Number analyzed (Participants) | 32 | 34
hours
  Day 15 | 3.5 (1.5) | 0 (0)
  Day 30 | 3.2 (1.0) | 3.1 (1.3)

15. Primary Outcome: Tmax of Venlafaxine Hydrochloride
Time Frame: Day 15 and Day 30 (24 hour sampling)
Population: PAS
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | LDX + Venlafaxine XR | Venlafaxine XR + LDX
Number analyzed (Participants) | 32 | 34
hours
  Day 15 | 0 (0) | 6.4 (0.8)
  Day 30 | 6.0 (1.3) | 5.9 (0.6)

16. Primary Outcome: Tmax of o-Desmethylvenlafaxine
Time Frame: Day 15 and Day 30 (24 hour sampling)
Population: PAS
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | LDX + Venlafaxine XR | Venlafaxine XR + LDX
Number analyzed (Participants) | 32 | 34
hours
  Day 15 | 0 (0) | 7.9 (1.2)
  Day 30 | 8.5 (1.7) | 7.9 (1.3)

17. Primary Outcome: Tmax of Composite (Venlafaxine + o-Desmethylvenlafaxine)
Time Frame: Day 15 and Day 30 (24 hour sampling)
Population: PAS
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | LDX + Venlafaxine XR | Venlafaxine XR + LDX
Number analyzed (Participants) | 32 | 34
hours
  Day 15 | 0 (0) | 7.3 (1.1)
  Day 30 | 7.1 (1.4) | 7.0 (1.2)

18. Secondary Outcome: Pulse Rate
Time Frame: Baseline and up to 39 days
Population: SAS
Measure: Mean (Standard Deviation); unit: bpm
Arm/Group | LDX + Venlafaxine XR | Venlafaxine XR + LDX
Number analyzed (Participants) | 40 | 37
bpm
  Baseline | 66.24 (7.940) | 66.55 (10.318)
  Up to 39 Days | 77.47 (8.621) | 81.72 (7.068)

ADVERSE EVENTS:
Groups:
- LDX (SPD489): Titration dosing period
- LDX + Venlafaxine XR/Venlafaxine XR + LDX: Combination dosing periods
- Venlafaxine XR Titration: Titration dosing period (Effexor XR 75, 150, and 225 mg)
- Venlafaxine XR Tapering: Tapering dosing period (Effexor XR 150 and 75 mg)
Arm/Group | LDX (SPD489) | LDX + Venlafaxine XR/Venlafaxine XR + LDX | Venlafaxine XR Titration | Venlafaxine XR Tapering
Serious Adverse Events (participants affected / at risk) | 1/40 | 0/67 | 0/37 | 0/67
Other Adverse Events (participants affected / at risk) | 33/40 | 46/67 | 25/37 | 20/67
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LDX (SPD489) (N=40) | LDX + Venlafaxine XR/Venlafaxine XR + LDX (N=67) | Venlafaxine XR Titration (N=37) | Venlafaxine XR Tapering (N=67)
Presyncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LDX (SPD489) (N=40) | LDX + Venlafaxine XR/Venlafaxine XR + LDX (N=67) | Venlafaxine XR Titration (N=37) | Venlafaxine XR Tapering (N=67)
Palpitations (Cardiac disorders) | 8 (11) | 2 (3) | 0 (0) | 0 (0)
Vision Blurred (Eye disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 3 (3) | 11 (14) | 3 (3) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 2 (3) | 2 (2) | 3 (3) | 2 (2)
Dry Mouth (Gastrointestinal disorders) | 10 (13) | 6 (6) | 7 (8) | 0 (0)
Nausea (Gastrointestinal disorders) | 6 (7) | 4 (4) | 7 (9) | 6 (7)
Stomach Discomfort (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Chest Pain (General disorders) | 3 (3) | 1 (1) | 0 (0) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 12 (21) | 0 (0) | 9 (10) | 0 (0)
Back Pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 3 (3) | 7 (9) | 4 (5) | 7 (7)
Headache (Nervous system disorders) | 7 (8) | 13 (17) | 6 (6) | 3 (3)
Somnolence (Nervous system disorders) | 7 (7) | 0 (0) | 7 (7) | 3 (3)
Anxiety (Psychiatric disorders) | 5 (7) | 2 (2) | 0 (0) | 0 (0)
Euphoric Mood (Psychiatric disorders) | 3 (4) | 0 (0) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 7 (7) | 5 (6) | 3 (5) | 0 (0)
Urinary Hesitation (Renal and urinary disorders) | 0 (0) | 5 (5) | 0 (0) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 5 (5) | 0 (0) | 0 (0)
Libido Decreased (Psychiatric disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If a multicenter publication is not submitted within twelve (12) months after conclusion, abandonment or termination of the Study at all sites, or after Sponsor confirms there shall be no multicenter Study publication, the Institution and/or such Principal Investigator may publish the results from the Institution site individually.